CLINICAL TRIAL: NCT05970549
Title: DIVE: Deployment of Irrigating Intraventricular Catheter System for Intraventricular Hemorrhage
Brief Title: Intraventricular Catheter System for IVH
Acronym: DIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: IRRAS (Industry)
Responsible Party: Principal Investigator, Christopher P Kellner, Assistant Professor in Neurosurgery, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01815
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Intraventricular Hemorrhage (IVH)

STUDY DESIGN:
Intervention Model Description: The IRRAflow® System is an active fluid exchange system in which intracranial pressure (ICP) monitoring, active controlled irrigation and passive drainage are combined in one system. The system consists of 3 items; control unit (i) and two sterile disposable parts: (ii) Intelligent Digital Cassette (Tube Set) and (iii) dual-lumen Catheter.
Masking Description: There will be no masking involved. The proposed study is a single center retrospective and prospective cohort, controlled, single-center, phase 1 study evaluating the safety and radiographic outcomes associated use of the IRRAS catheter compared to standard of care external ventricular drains.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- IRRAflow with Active Fluid Exchange arm (Experimental): The analysis of the IRRAS catheter will occur prospectively if it is determined the patient meets the enrollment criteria.
  Interventions: Device: IRRAflow® Active Fluid Exchange System; Procedure: Non-contrast head CTs
- Retrospective analysis of traditional external ventricular drains (Active Comparator): The retrospective analysis will be performed on the last 60 traditional external ventricular drains.
  Interventions: Device: Traditional extraventricular drain

INTERVENTIONS:
Device: IRRAflow® Active Fluid Exchange System — All patients in the prospective arm of the study who met the study criteria and consent will be enrolled in the IRRAflow with Active Fluid Exchange arm.
  Insertion of the IRRaflow catheter will be performed by neurosurgical attendings and residents who are privileged to place external ventricular drains and who have be instructed on how to appropriately connect the inserted IRRAflow catheter to the system. The on-site IRRAflow instructor will be present and available at all time to assist with any issues or questions should they arise.
  Other Names: IRRAflow® CNS System
  Arms: IRRAflow with Active Fluid Exchange arm
Device: Traditional extraventricular drain — The retrospective analysis will be performed on the last 60 traditional external ventricular drains.
  Arms: Retrospective analysis of traditional external ventricular drains
Procedure: Non-contrast head CTs — Non-contrast head CTs will be performed at least every 48 hours to document effectiveness. This frequency is standard, if not more frequent as necessary, for patients with external ventricular drainage and intraventricular hemorrhage. Scans are routinely obtained at this frequency to evaluate, for example: evacuation of hemorrhage, admission pathology, post-placement of catheters, any change in neurological exam, or after elevations in intracranial pressure. With these common CT scans we will be able to assess the efficacy of the IRRAflow catheter on the specified parameters. These scans are routinely performed due to this pathology and as such are covered as a necessity of the hospitalization by the insurance companies. MRI may be used in place of a CT scan if medically indicated as determined by the neurosurgical attending or neurocritical care attending according to standard of care for treatment of the neurological pathology.
  Arms: IRRAflow with Active Fluid Exchange arm

SUMMARY:
The purpose of this research study is to evaluate the safety and outcomes associated with the use of IRRAflow® System catheters in externally draining intracranial fluid to reduce intracranial pressure. This study will be comparing the IRRAflow® system to standard of care catheters used in the same procedure. The IRRAflow® system is FDA approved for this procedure.

DETAILED DESCRIPTION:
Intracranial hemorrhagic conditions can rapidly cause brain damage and often considered life- threatening. Of these, Intracerebral hemorrhagic (ICH) is the most common type of hemorrhagic stroke and is associated with higher rates of morbidity and mortality than all stroke subtypes.

Management of hemorrhagic patients is typically orchestrated by neurosurgeons and neuro-intensivists. Comprehensive care should include surveillance and monitoring of Intra Cranial Pressure (ICP), Cerebral Perfusion Pressure (CPP), and hemodynamic function. Furthermore, prevention of infection, complications of immobility through positioning and mobilization within physiological tolerance play an important role in optimizing outcomes after ICH.

There are multiple approaches to facilitating Cerebrospinal Fluid (CSF) drainage and monitor ICP. Routinely, intracranial pressure is measured by use of devices inserted into the brain parenchyma or cerebral ventricles. A Ventricular Catheter (VC) inserted into the lateral ventricle allows for drainage of CSF to help reduce ICP. Although CSF drainage is a vital sequence in patient management, there are reported risks including infection and limitations related to erroneous readings associated with current ICP monitors. Physicians lack the appropriate tools to employ active intermittent aspiration and drainage with continuous ICP monitoring.

The current clinical study is being initiated to evaluate the hypothesis that active irrigation by IRRAflow will reduce the time needed for clearance of intraventricular blood from intraventricular space.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years of age
* Intraventricular hemorrhage documented on head CT or MRI scan
* Need of cerebrospinal fluid drainage
* Indication for active treatment evaluated by the treating physicians
* Signed informed consent obtained by patient or Legal Authorized Representative
* Treatment possible within 72 hours of ictus

Exclusion Criteria:

* Patient has fixed and dilated pupils
* Pregnant or nursing women (fertile female participants will be required to take a validated pregnancy test for evaluation of pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Residual blood volume | At day 5
  Residual blood volume on post bleed day 5

SECONDARY OUTCOMES:
Serious adverse events | up to 48 hours post-procedure
  Number of serious adverse events
Hospital quality metrics | up to 48 hours post-procedure
  Length of stay in the NSICU as a quality metrics
Length of stay in the NSICU | up to 48 hours post-procedure
  Length of hospital stay in the as a quality metrics
Direct hospitalization costs | up to 48 hours post-procedure
  Direct hospitalization costs

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Kellner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
In order to minimize any privacy risks to the patients participating, IPD data will not be shared.